CLINICAL TRIAL: NCT06697691
Title: Construction of a Clinical Prediction Model for In-Hospital Rebleeding in Patients With Acute Non-Venous Upper Gastrointestinal Bleeding
Brief Title: Clinical Prediction Model for In-Hospital Rebleeding in Acute Non-Variceal Upper Gastrointestinal Bleeding
Status: Recruiting | Type: Observational
Sponsor: Junwei Yan (Other)
Responsible Party: Sponsor-Investigator, Junwei Yan, Principal Investigator, Wuhan Central Hospital
Organization: Wuhan Central Hospital (Other)
Other Study IDs: ANVUGIB-2024-001
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Acute Non-variceal Upper Gastrointestinal Bleeding
Keywords: rebleeding; acute non-variceal upper gastrointestinal bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ANVUGIB is a serious condition that can cause symptoms like vomiting blood or passing black stools. Although treatments have improved, about 10% to 30% of patients experience rebleeding shortly after their initial treatment, which increases the risk of death.

Currently, doctors use tools like the Glasgow-Blatchford Score, Rockall Score, and AIM65 Score to predict how patients with ANVUGIB might recover. However, these tools are not very effective at identifying patients who are at risk for rebleeding. This study aims to create a new, more accurate prediction model to help doctors identify high-risk patients earlier. The investigators believe that a new predictive model, which combines patient symptoms, lab test results, and imaging findings, will improve the ability to identify patients at high risk of rebleeding compared to existing tools.The goal is to provide doctors with a more reliable tool to guide their decisions, such as when to give preventive treatments or increase monitoring. This could lead to better outcomes and reduce the risk of complications or death.

This study uses patient data collected during routine care to develop and test the new model, ensuring the findings are directly applicable to real-world clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* age exceeding 18 years,
* Clinical diagnosis of Acute Non-Variceal Upper Gastrointestinal Bleeding ,
* patients who underwent endoscopy within 24 hours of admission with confirmation of non-variceal bleeding

Exclusion Criteria:

* Upper Gastrointestinal Bleeding during hospitalization;
* transfer from other hospitals;
* variceal bleeding;
* lower gastrointestinal bleeding.;
* bleeding attributed to systemic diseases like disseminated intravascular coagulation (DIC) and hematological disorders;
* patients with incomplete clinical data or laboratory test results;
* patients who either requested early discharge or declined gastroscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients hospitalized for AUGIB at the Central Hospital of Wuhan from December 2021 to December 2023
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
relbeeding | up to 7 days
  Rebleeding was defined as hematemesis, hematochezia, and/or melena within 7 days of the initial bleeding, accompanied by hemodynamic instability or a decrease in hemoglobin of at least 2 g/dl within 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- the Central Hospital of Wuhan, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided